CLINICAL TRIAL: NCT02255825
Title: Development of an Optimal Approach to Return of Results for Families Undergoing Next-generation Sequencing for Prenatal Diagnosis.
Brief Title: Development of an Optimal Approach to Return of Results for Next-generation Sequencing for Prenatal Diagnosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting verification of assay
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Louise Laurent, MD/PhD, MD/PhD, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 140456
Record Dates: First submitted 2014-09-24; First posted 2014-10-03 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Major Fetal Anomaly
MeSH Terms: interventions — Whole Genome Sequencing; Amniocentesis; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Amniocentesis will be performed, Whole Genome Sequencing will not be performed, and psychosocial assessment will be performed.
  Interventions: Procedure: Amniocentesis; Other: Psychosocial assessment
- Intervention Group (Experimental): Amniocentesis will be performed, Whole Genome Sequencing will be performed if the karyotype is normal, and psychosocial assessment will be performed.
  Interventions: Genetic: Whole Genome Sequencing; Procedure: Amniocentesis; Other: Psychosocial assessment

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Whole genome sequencing in a CLIA lab and return of results.
  Arms: Intervention Group
Procedure: Amniocentesis — Note: this is being performed on all subjects as a clinical (not research) procedure
Other: Psychosocial assessment — Use of EPDS and STAI for assessment of maternal and paternal mood

SUMMARY:
To gain knowledge about how patients undergoing prenatal diagnosis for a fetal abnormality understand and react to Whole Genome Sequencing (WGS) testing, so that the investigators can develop more ethical and responsible approach to patient education, counseling, and return of results for patients.

DETAILED DESCRIPTION:
Although whole exome sequencing (WES) was first used for identification of the genetic cause of a disease only in 2009 and whole genome sequencing (WGS) in 2010, and questions remain about their performance as clinical tests, they are already being offered to patients and doctors as a clinical test by several laboratories certified by the US government (14 labs for WES and 5 labs for WGS). The results from WES and WGS can be complex and confusing, even for doctors and scientists who work with this technology on a daily basis; for patients, the process of deciding whether to have WES or WGS testing, undergoing the testing, receiving the results, and trying to use the results for further decision-making could be quite stressful. Currently, this process occurs in an unstandardized fashion, with some patients receiving extensive education and counseling, and others receiving almost none. There is a critical need to identify patient needs and desires in this area, and to develop strategies to satisfy them. The primary goal of this project is to gain knowledge about how patients undergoing prenatal diagnosis for a fetal abnormality understand and react to WGS testing, so that we can develop a more ethical and responsible approach to patient education, counseling, and return of results for patients . In order to do this, we need to evaluate parents' understanding of the utility and limitations of the technology, parents' preferences regarding the types of results they want to receive, and the psychological impact of receiving results from this technology. We will enroll 30 families consisting of a woman carrying a fetus with a major abnormality identified by ultrasound, and the father of the fetus, who have opted for amniocentesis for standard prenatal diagnostic testing (karyotyping, fluorescence in situ hybridization (FISH) and/or microarray testing). Half of the families will serve as controls, who will only have standard prenatal diagnostic testing. For the other half of the families, WGS will be performed in addition to standard diagnostic testing. For all 30 cases, we will perform psychosocial evaluations (including assessments of the subjects' mood, understanding of the technology and preferences for return of results) at the time of enrollment, at the time of return of CLIA-certified genetic testing results (karyotype, FISH, microarray, and/or WGS), and after completion of the pregnancy. In this way, we will learn whether participants are receiving adequate education about next-generation sequencing to make informed choices, what the range of preferences are for return of results in a prenatal population (and whether this changes when new methods for prenatal diagnosis are employed), and whether the use of WGS imposes additional psychological stress compared to standard prenatal diagnostic tests. This study will be carried out in a stepwise and carefully monitored environment, with progress overseen by an Independent Data Monitoring Committee in order to maximize the knowledge gained while minimizing potential harms.

ELIGIBILITY:
Inclusion Criteria:

* Subject(s) 18 years or older (both mom and father of baby (FOB)
* Subject is undergoing prenatal testing for a major fetal anomaly

Exclusion Criteria:

* Mothers or fathers of the affected fetus are under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Change in maternal mood (focused on assessment of depression) | At enrollment and 3 months after completion of pregnancy (expected to be 8 months after enrollment)
  Compare mood measured by EPDS between enrollment and 3 months after completion of pregnancy
Change in paternal mood (focused on assessment of depression) | At enrollment and 3 months after completion of pregnancy (expected to be 8 months after enrollment)
  Compare mood measured by EPDS between enrollment and 3 months after completion of pregnancy

SECONDARY OUTCOMES:
Change in maternal mood (focused on assessment of anxiety) | At enrollment and 3 months after completion of pregnancy (expected to be 8 months after enrollment)
  Compare anxiety measured by STAI between enrollment and 3 months after completion of pregnancy
Change in paternal mood (focused on assessment of anxiety) | At enrollment and 3 months after completion of pregnancy (expected to be 8 months after enrollment)
  Compare anxiety measured by STAI between enrollment and 3 months after completion of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Health Sciences, Fetal Care and Genetics, San Diego, California, United States